CLINICAL TRIAL: NCT05291260
Title: MUlticenter Randomized Controlled Trial on Nonoperative Versus Operative Treatment for Acute Complete tearS of the Ulnar Collateral ligAment of the Thumb: Cost- Effectiveness and Functional Outcomes.
Brief Title: RCT on Nonoperative Versus Operative Treatment for Acute Complete tearS of the Ulnar Collateral ligAment of the Thumb
Acronym: MUSCAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonessenhuis, Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78886.100.21
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-09

CONDITIONS: Ulnar Collateral Ligament Sprain; Skier's Thumb
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Masking Description: Not possible for surgical intervention vs cast immobilization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cast immobilization (Experimental): Cast immobilization to immobilize the thumb for 4 weeks. After 2 weeks the thumb will be re-examined to determine if surgery is required. It is expected that at re-evaluation at 2 weeks after starting the cast treatment about 1 in 10 patients will still need surgery.
  Interventions: Procedure: Cast immobilization
- Surgery (Active Comparator): The intervention is compared to surgery, which is standard treatment for complete ulnar collateral ligament ruptures.
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Cast immobilization — A cast to immobilize the MCP, in 10-30 degrees (slight) flexion (neutral position), and the CMC joint, in 30-40 degrees palmar abduction, is applied (IP joint is free).
  Arms: Cast immobilization
Procedure: Surgical treatment — In general, two surgical techniques are described in literature and used in daily clinical practice:
  * If the UCL is ruptured in the middle of the ligament, sutures are used to reattach the ligament remnants together.
  * When no viable UCL ligaments are present, the UCL is reattached directly to the bone using suture anchors.
  Arms: Surgery

SUMMARY:
A complete rupture of the ulnar collateral ligament (UCL) of the thumb must heal in order to regain proper function of the thumb. Guidelines recommend surgery for complete UCL ruptures, including Stener lesions. This recommendation is based on expert opinion, anatomic theories and low quality retrospective case series. High quality studies comparing cast immobilization with operative treatment are lacking. Research has shown that in about 9 out of 10 patients, a complete UCL rupture, including Stener Lesions, can also be treated with a cast alone for 6 weeks and no surgery is needed. We hypothesize that cast immobilization is non-inferior regarding functional outcome and carries concomitant lower costs compared with operative treatment for complete UCL ruptures, including Stener Lesions.

The project aims to conduct a multicenter randomized controlled trial and cost-effectiveness analysis comparing operative and nonoperative treatment for complete UCL ruptures, including Stener Lesions. The project will take four years, from preparation to reporting of the results. In the following years, implementation will be achieved in collaboration with the Dutch hand surgery committees (NVvH and NVPC), health insurance companies, and medical experts.

Research question Is nonoperative treatment with splint immobilization non-inferior to immediate operative treatment regarding functional outcome and does it lead to lower costs in adult patients with an acute complete UCL rupture, including Stener Lesions?

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Dutch or English speaking patients
* Patients with an acute complete UCL rupture, with or without a Stener Lesion, diagnosed using physical examination, performed by the hand surgeon. When providing radically directed force to the proximal phalanx (radial deviation stress) as the thumb metacarpal is stabilized, criteria 1 AND 2 must be present to confirm the diagnosis of a complete UCL rupture:

  * no firm endpoint in the MCP joint AND
  * at least more than 35 degrees of laxity in the MCP joint (measured with the MCP joint in extension or in 30 degrees of flexion) OR more than 15 degrees difference in laxity compared with the uninjured side.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Michigan Hand outcome Questionnaire (MHQ) | 6 months
  The MHQ, expressed as the MHQ at 6 months (from randomization to 6 months after) is the primary endpoint of the study. The MHQ is a validated tool for assessment of functional outcome in patients with pathology of the hand. The MHQ is a questionnaire divided in six subscales; overall hand function, activities of daily living (ADLs), pain, work performance, aesthetics and patient satisfaction with hand function. Each subscale has a formula to calculate a score. The final score is a summation of the six individual item-scores divided by six and goes from 0 (severe disability) to 100 (no disability).

SECONDARY OUTCOMES:
Patient-Specific Functional Scale (PSFS) | at randomization, 2, 3, 6 and 12 months after randomization.
  a self-reported, patient-specific outcome measure, designed to assess functional change, primarily in patients presenting with musculoskeletal disorders. Patients are asked to identify up to five important activities they are unable to perform or are having difficulty with as a result of their problem i.e. putting socks on. In addition to identifying the activities, patients are asked to rate, on an 11-point scale, the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified and are given the chance to nominate new problematic activities that might have arisen during that time. "0" represents unable to perform, "10" represents able to perform. Patients select a value that best describes their current level of ability on each activity assessed.
EQ-5D-5L | at randomization, 2, 3, 6 and 12 months after randomization.
  a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgment. The score on the five dimensions can be presented as a health profile or can be converted into a utility score based on an available Dutch scoring algorithm (www.euroqol.org). The area under the curve of utility scores over time will be used to express the effect on quality of life in QALY's.
Michigan Hand outcome Questionnaire (MHQ) | at randomization, 2, 3 and 12 months after randomization.
  see above
The Numeric Pain Rating Scale (NPRS) | at randomization, 2, 3, 6 and 12 months after randomization.
  will be used to assess pain, where 0 implies no pain and 10 the worst possible pain measured
Patient satisfaction | at randomization, 2, 3, 6 and 12 months after randomization.
  will be measured by using the ICHOM Satisfaction with treatment results questionnaire (self designed by ICHOM)
The adapted Dutch institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ) | at 2 months (over the last 2 months), 3 (over the last month), 6 (over the last 3 months), and 12 (over the last 3 months) months after randomization
  to measure the amount of medical consumption due to a complete tear of the UCL (the questionnaire is adjusted for this study)
Range of motion (ROM) | 4 weeks, 3, 6 and 12 months after randomization.
  flexion and extension of the metacarpophalangeal (MCP) joint and interphalangeal joint (IP) and palmar abduction of the carpometacarpal (CMC) joint are measured with a goniometer. The first measurement is performed at both sides.
Kapandji-score | 4 weeks, 3, 6 and 12 months after randomization.
  assessing the opposition of the CMC joint. The opposition test consists of touching the four long fingers with the tip of the thumb. The more the tip of the thumb is able to oppose to the base of the pink, the higher the score will be.
Complications | 4 weeks, 3, 6 and 12 months after randomization.
  * Conservative treatment: pressure ulcers, neuropraxia or injury to the sensory superficial branches of radial nerve, arthrosis, chronic instability or limited function.
  * Perioperative: vascular damage, nerve or tendon laceration.
  * Postoperative: surgical site infection, repeat operation, pressure ulcers, neuropraxia or injury to the sensory superficial branches of radial nerve, arthrosis, chronic instability or limited function.
  Peri- and postoperative complications will be recorded according tot the Clavien-Dindo Classification for hand surgery. Repeat operation and subsequent description of the additional treatment method will be reported.
The adapted Dutch institute for Medical Technology Assessment (iMTA)Productivity Cost Questionnaire (iPCQ) | at 2 months (over the last 2 months), 3 (over the last month), 6 (over the last 3 months), and 12 (over the last 3 months) months after randomization
  to measure the amount sick leave from work or lost productivity while at work and out-of pocket expenses due to a complete tear of the UCL and the questionnaire is adjusted for this study.
Grip strength | 4 weeks, 3, 6 and 12 months after randomization.
  measured with a hand-held dynamometer. The measurement includes three trials of maximum grip force using the second handle of a calibrated dynamometer, with the elbow in 90° flexion. Dynamometer settings will be based on patients' hand size. Each center will use the same type of dynamometer. The mean score of three trials will be used for analysis as an absolute measure. The first measurement is performed at both sides.
Pinch strength | 4 weeks, 3, 6 and 12 months after randomization.
  key pinch/lateral pinch and tip pinch will be measured. Key pinch includes three trials of maximum force between the radial side of the index finger and the pulp of the thumb, using a calibrated pinch gauge, with the elbow in 90° flexion. Tip pinch includes three trials of maximum force between the tip of the index finger and the tip of the thumb, using a calibrated pinch gauge, with the elbow in 90° flexion. Each center will use the same type of pinch gauge. The mean score of three trials will be used for analysis as an absolute measure. The first measurement is performed at both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Mark van Heijl, MD, PhD, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
An official Data Management Plan has been developed, in accordance with the official format used in the Netherlands.
Supporting Information: Study Protocol
Time Frame: When the manuscripts are published
URL: https://muscatstudie.nl/

REFERENCES:
- [Background] Pulos N, Shin AY. Treatment of Ulnar Collateral Ligament Injuries of the Thumb: A Critical Analysis Review. JBJS Rev. 2017 Feb 21;5(2):e3. doi: 10.2106/JBJS.RVW.16.00051. No abstract available. PMID 28248741
- [Background] Pichora DR, McMurtry RY, Bell MJ. Gamekeepers thumb: a prospective study of functional bracing. J Hand Surg Am. 1989 May;14(3):567-73. doi: 10.1016/s0363-5023(89)80026-7. PMID 2738347
- [Background] Landsman JC, Seitz WH Jr, Froimson AI, Leb RB, Bachner EJ. Splint immobilization of gamekeeper's thumb. Orthopedics. 1995 Dec;18(12):1161-5. doi: 10.3928/0147-7447-19951201-06. PMID 8749294
- [Background] Samora JB, Harris JD, Griesser MJ, Ruff ME, Awan HM. Outcomes after injury to the thumb ulnar collateral ligament--a systematic review. Clin J Sport Med. 2013 Jul;23(4):247-54. doi: 10.1097/JSM.0b013e318289c6ff. PMID 23615487
- [Background] Mikhail M, Wormald JCR, Thurley N, Riley N, Dean BJF. Therapeutic interventions for acute complete ruptures of the ulnar collateral ligament of the thumb: a systematic review. F1000Res. 2018 Jun 8;7:714. doi: 10.12688/f1000research.15065.1. eCollection 2018. PMID 30057756
- [Derived] de Haas L, van Hoorn B, van de Lucht V, Schep N, Dijkgraaf M, van Heijl M; MUSCAT Trial Collaborator group. Study protocol for a multicenter non-inferiority randomized controlled trial to assess functional outcomes and cost-effectiveness of a primarily non-operative treatment strategy with cast immobilization versus immediate operative treatment followed by cast immobilization for patients with complete ulnar collateral ligament ruptures, including Stener lesions: MUSCAT study. Trials. 2024 Oct 28;25(1):723. doi: 10.1186/s13063-024-08576-x. PMID 39468632